CLINICAL TRIAL: NCT07210827
Title: The Effect of Nasal Septal Deviation on Maxillary Sinus Volumes and Development of Maxillary Sinusitis :A CT Study.
Brief Title: Deviated Nasal Septum Effect on Maxillary Sinus Volumes and Development of Maxillary Sinusitis by CT
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Rana Emad Ali, Ent resident, Assiut University
Other Study IDs: CT in nasal septal deviation
Record Dates: First submitted 2025-09-30; First posted 2025-10-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: Deviated Nasal Septum and Maxillary Sinusitis
MeSH Terms: conditions — Maxillary Sinusitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
By using CT of the nose and paranasal sinuses, we'll study the effect of nasal septum deviation on maxillary sinus volumes, assess the association between the severity and type of nasal septum deviation and the occurrence of maxillary sinusitis and compare the maxillary sinus volume on the deviated side with that of the contralateral side.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years.
2. Availability of high-resolution CT scans of paranasal Sinuses (axial, coronal, sagittal views).
3. Adequate imaging quality allowing sinus volumetry and septal deviation measurement.
4. Anatomical landmarks visible: Crista galli, hard palate, choanae, uncinate process/OMC region clearly identifiable to permit NSD measurement and sinus segmentation.

Exclusion Criteria:

1. Age < 18 years.
2. Previous sinonasal or maxillofacial surgery.
3. History of facial trauma or fractures affecting the nasal septum or sinus walls.
4. Sinonasal tumors, polyps, or large cysts.
5. Congenital craniofacial anomalies (e.g., cleft palate).
6. head and neck syndromes.
7. Cases with systemic diseases affecting growth and development.

   -

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients presented to outpatient clinic at Assiut University hospital complaining of nasal symptoms like nasal obstruction, rhinorrhea ,headache, and recurrent sinusitis.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
CT based comparison in cases with deviated nasal septum | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Abdelaleem, Study Chair — Professor at ENT department,Assiut University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Razavi M, Shams N, Pirasteh SMA. Determining the effects of deviated nasal septum on maxillary sinus volume using cone-beam computed tomography. Immunopathol Persa. 2023;9(1):e34427
- [Background] Elahi MM, Frenkiel S, Fageeh N. Paraseptal structural changes and chronic sinus disease in relation to the deviated septum. J Otolaryngol. 1997 Aug;26(4):236-40. PMID 9263892
- [Background] Serifoglu I, Oz II, Damar M, Buyukuysal MC, Tosun A, Tokgoz O. Relationship between the degree and direction of nasal septum deviation and nasal bone morphology. Head Face Med. 2017 Feb 28;13(1):3. doi: 10.1186/s13005-017-0136-2. PMID 28245851